CLINICAL TRIAL: NCT05944575
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Ventricular Rate Control in Patients With Persistent Atrial Fibrillation
Brief Title: Effect of taVNS on Heart Rate in Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Burrell College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Harald Stauss MD PhD, Professor of Pharmacology, Burrell College of Osteopathic Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0104_2022
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: vagus nerve stimulation; Electrocardiogram; Heart rate
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Treatment for each patient will crossover (after one week) from an active taVNS to an inactive sham-taVNS treatment or vice versa (depending on randomization).
Who Masked: Participant
Masking Description: Participants will not be told if the location of the clip electrode will be for active taVNS or for sham-taVNS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Intervention (Active Comparator): Participants will self-administer active taVNS for 30 min per day for 7 days.
  Interventions: Device: active taVNS
- Sham Intervention (Sham Comparator): Participants will self-administer sham-taVNS for 30 min per day for 7 days.
  Interventions: Device: sham-taVNS

INTERVENTIONS:
Device: active taVNS — The clip electrode will be attached to the cymba conchae of the left ear, the location of the auricular branch of the vagus nerve.
  Arms: Active Intervention
Device: sham-taVNS — The clip electrode will be attached to the lobule of the left ear that is not innervated by the auricular branch of the vagus nerve.
  Arms: Sham Intervention

SUMMARY:
The goal of this clinical trial is to investigate the effects of non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) in patients with persistent atrial fibrillation. taVNS is a treatment through which a small electrical current is applied to a specific location of the left ear. The main question to answer is whether taVNS will reduce the heart rate in patients with persistent atrial fibrillation. After appropriate training, participants will self-administer taVNS for 30 minutes every day for two weeks. During one of the two weeks (randomized order), the clip electrode, delivering the electrical current will be attached to the cymba conchae of the left ear, while during the other week the clip electrode will be attached to the lobule of the left ear. During both weeks, the electrocardiogram (ECG) will be monitored continuously through a small ECG patch that is placed on the chest. Participants will meet with the investigators at the beginning of the study, after 7 days and at the end of the study (after 14 days). Researchers will compare the ECG obtained during the two weeks and evaluate if the heart rate differs between the two study weeks.

DETAILED DESCRIPTION:
In a previous study (Dalgleish et al., 2021), the investigators found that taVNS lengthens the PQ-interval in healthy study participants with regular sinus rhythm. This finding indicates that taVNS slows AV-conduction. Thus, it is reasonable to assume that taVNS may lower ventricular rate in patients with persistent atrial fibrillation. This assumption is in line with a recent study (Stavarakis et al., 2020) demonstrating reduced atrial fibrillation burden in patients with paroxysmal atrial fibrillation in response to a 6-month taVNS intervention.

The investigators hypothesize that taVNS reduces ventricular rate in patients with persistent atrial fibrillation. This hypothesis is based on the finding that taVNS lengthens the PQ-interval in healthy individuals with sinus rhythm (Dalgleish et al., 2021), demonstrating that taVNS slows AV-nodal conduction. Thus, it is conceivable that taVNS reduces the number of atrial excitations that are transmitted into the ventricles in patients with persistent atrial fibrillation. This effect should result in a lower ventricular rate. Testing this hypothesis is significant, because if the hypothesis would be verified, taVNS would have the potential to elicit an additive effect to AV-nodal blocking agents, and thus, may allow to reduce the dose of such drugs, effectively reducing potential adverse effects.

The study is designed as a two-week randomized cross-over study. Participants will start with either taVNS or sham-taVNS (randomly assigned) during the first week and then switch to the other intervention during the second week of the study. Throughout the two-week study, ambulatory ECG will be recorded using an ECG patch that allows continuous ECG recording for up to 14 days. Participants will self-apply taVNS or sham-taVNS for 30 min every day throughout the 2-week study.

Participants will meet with the investigators 3 times throughout the 2-week study protocol: On the first study day, participants will be instrumented with the ECG patch and instructed in the use of the taVNS device. In addition, patients will be instructed to keep a diary to record the time of the taVNS/sham-taVNS application, the stimulation parameters, and any potential therapeutic or adverse effects. The second study visit will occur at the end of the first study week. During this meeting, the function of the ECG patch and taVNS device will be verified, the diary will be inspected to verify protocol adherence, and the intervention will be switched to either taVNS or sham-taVNS application (depending on randomization). The final study visit will occur at the end of the study (after 2 weeks). The ECG patch will be retrieved, and the diary inspected for protocol adherence.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Persistent atrial fibrillation
* On anti-coagulation throughout the study

Exclusion Criteria:

* Below 18 years of age
* Pregnancy
* Signs or history of vestibulocochlear neuronitis or nerve damage (e.g., hearing loss or tinnitus)
* Signs or history of epilepsy
* Not on anti-coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Weekly ventricular rate | After one week of treatment or sham treatment
  The average ventricular rate (obtained from the ECG patch) during the week with active taVNS (active intervention arm) will be compared with the average ventricular rate during the week with sham-taVNS (sham intervention arm).
Ventricular rate during taVNS application | During 30 minutes of treatment or sham treatment
  The ventricular rate (obtained from the ECG patch) during the 30 min of taVNS application will be compared with the ventricular rate during the 30 min of sham-taVNS application for each of the 7 days of each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Harald M Stauss, MD, PhD, Principal Investigator — Burrell College of Osteopathic Medicine
Locations (1):
- Burrell College of Osteopathic Medicine, Las Cruces, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Dalgleish AS, Kania AM, Stauss HM, Jelen AZ. Occipitoatlantal decompression and noninvasive vagus nerve stimulation slow conduction velocity through the atrioventricular node in healthy participants. J Osteopath Med. 2021 Feb 18;121(4):349-359. doi: 10.1515/jom-2020-0213. PMID 33694346
- [Background] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678